CLINICAL TRIAL: NCT01256424
Title: A Randomized Phase II Dose-finding Study of Hexaminolevulinate (HAL) Photodynamic Therapy (PDT) in Patients With Low/Moderate-grade Cervical Intraepithelial Neoplasia (CIN1 or 2)
Brief Title: Dose-finding Study of Hexaminolevulinate (HAL) Photodynamic Therapy (PDT) to Treat Cervical Neoplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Photocure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PC CE203/10
Record Dates: First submitted 2010-12-07; First posted 2010-12-08 (Estimated); Results first posted 2014-08-21 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: CIN
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Lighting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- HAL 5% with illumination (Experimental): HAL PDT 5%
  Interventions: Drug: HAL 5% with illumination
- HAL 1% with illumination (Experimental): HAL PDT 1%
  Interventions: Drug: HAL 1% with illumination
- HAL 0.2% with illumination (Experimental): HAL PDT 0.2%
  Interventions: Drug: HAL 0.2% with illumination
- Placebo ointment without illumination (Placebo Comparator): Placebo without illumination
  Interventions: Drug: Placebo ointment without illumination

INTERVENTIONS:
Drug: HAL 5% with illumination — Treatment with a singe dose of 2g, HAL 5% ointment followed by photoactivation
  Arms: HAL 5% with illumination
Drug: HAL 1% with illumination — Treatment with a singe dose of 2g, HAL 1% ointment followed by photoactivation
  Arms: HAL 1% with illumination
Drug: HAL 0.2% with illumination — Treatment with a singe dose of 2g, HAL 0.2% ointment followed by photoactivation
  Arms: HAL 0.2% with illumination
Drug: Placebo ointment without illumination — Treatment with a singe dose of 2g placebo ointment, no photoactivation
  Arms: Placebo ointment without illumination

SUMMARY:
An effective and safe medical therapy would be most welcome to reduce the need for surgical interventions and related adverse events and psychological impact on patients with cervical cancer precursors. In this clinical trial, the investigators propose to evaluate the efficacy and safety of photodynamic therapy (PDT) using hexaminolevulinate (HAL) for mild to moderate-grade CIN (grade 1-2).

ELIGIBILITY:
Inclusion Criteria:

* Patients with ectocervical CIN1 or CIN2 as verified by local pathology (biopsy) obtained within the last month
* Satisfactory colposcopy examination including:

  * visibility of entire transformation zone including the squamocolumnar junction and
  * visibility of entire lesion margin
* Negative endocervical os by colposcopy
* Colposcopical visible lesion at visit 2, before treatment
* Patients with an average sized uterine cervix (approximately 27mm diameter) suitable for application of the Klemcap
* Age 18 or above
* Written informed consent signed

Exclusion Criteria:

* Previous treatment of CIN or invasive disease
* Lesion(s) extending to the vaginal vault
* Atypical glandular cells (AGC) or adenocarcinoma in situ (AIS) on cytology, malignant cells on cytology or histology or other suspicion of either micro-invasive or invasive disease
* Suspicion of endocervical disease on colposcopy
* Current severe pelvic inflammatory disease, severe cervicitis, or other severe gynaecological infection as per colposcopy and clinical examination
* Undiagnosed vaginal bleeding
* History of toxic shock syndrome
* Known or suspected porphyria
* Known allergy to hexaminolevulinate or similar compounds (e.g. methyl aminolevulinate or aminolevulinic acid)
* Pregnancy, or intention to become pregnant during the study period
* Nursing
* Childbirth or miscarriage within six weeks of enrolment
* Use of heart pacemaker
* Participation in other clinical studies either concurrently or within the last 30 days
* Risk of poor protocol compliance. Patient participation should be considered with respect to living far away from the hospital, plans for moving to another city/state, frequent travelling, planning to become pregnant, drug abuse/alcoholic, difficult working hours, family obligations, other illness (e.g. psychiatric), etc.
* Unwillingness to use adequate birth control (not abstinence) from screening until last PDT
* Patient is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2011-04; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hillemanns, MD, PhD, Principal Investigator — University Hospital Hannover
Locations (2):
- University Hospital Hannover, Hanover, Germany
- Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Derived] Hillemanns P, Garcia F, Petry KU, Dvorak V, Sadovsky O, Iversen OE, Einstein MH. A randomized study of hexaminolevulinate photodynamic therapy in patients with cervical intraepithelial neoplasia 1/2. Am J Obstet Gynecol. 2015 Apr;212(4):465.e1-7. doi: 10.1016/j.ajog.2014.10.1107. Epub 2014 Oct 31. PMID 25467012

RESULTS

PARTICIPANT FLOW:
Groups:
- HAL 5% With Illumination: Cervical PDT using Hexaminolevulinate: Treatment with a singe dose of 2g HAL 5% ointment followed by photoactivation
- HAL 1% With Illumination: Cervical PDT using Hexaminolevulinate: Treatment with a singe dose of 2g HAL 1% ointment followed by photoactivation
- HAL 0.2% With Illumination: Cervical PDT using Hexaminolevulinate: Treatment with a singe dose of 2g HAL 0.2% ointment followed by photoactivation
Period: Overall Study
Arm/Group | HAL 5% With Illumination | HAL 1% With Illumination | HAL 0.2% With Illumination | Placebo Ointment Without Illumination
Started | 65 | 67 | 62 | 68
Completed | 56 | 59 | 55 | 61
Not Completed | 9 | 8 | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Placebo Ointment Without Illumination: Cervical PDT using Hexaminolevulinate: Treatment with a singe dose of 2g placebo ointment, no photoactivation
- Total: Total of all reporting groups
Arm/Group | HAL 5% With Illumination | HAL 1% With Illumination | HAL 0.2% With Illumination | Placebo Ointment Without Illumination | Total
Number analyzed (Participants) | 65 | 67 | 62 | 68 | 262
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 65 | 67 | 62 | 68 | 262
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 67 | 62 | 68 | 262
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 0 | 4
  White | 64 | 65 | 61 | 68 | 258
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Lesion Response Rates of Three Different Doses of HAL PDT and Placebo at 3 Months After Treatment.
Description: Lesion response was defined by three variables: Histology, cytology and HPV. Patient response at three months required histology regression to CIN1 or normal, cytology of LSIL or less severe, and HPV negative.
Time Frame: 3 months after last treatment
Population: Patients with CIN2 at baseline, based on central histology review
Measure: Number; unit: percentage of patients
Arm/Group | HAL 5% With Illumination | HAL 1% With Illumination | HAL 0.2% With Illumination | Placebo Ointment Without Illumination
Number analyzed (Participants) | 19 | 29 | 19 | 21
percentage of patients | 95 | 69 | 63 | 57

2. Secondary Outcome: Comparison of HPV Response of Three Different Doses of HAL PDT and Placebo at 3 Months After Treatment.
Description: HPV response was defined as clearance of baseline HPV infection, asssessed by genotype
Time Frame: 3 months after treatment
Population: Patients with CIN2 at baseline, based on central histology read, and HPV positive at baseline
Measure: Number; unit: percentage of patients
Groups:
- Placebo Ointment Without Illumination: Cervical PDT using Hexaminolevulinate: Treatment with a singe dose of 2g placebo ointment,no photoactivation
Arm/Group | HAL 5% With Illumination | HAL 1% With Illumination | HAL 0.2% With Illumination | Placebo Ointment Without Illumination
Number analyzed (Participants) | 13 | 24 | 17 | 18
percentage of patients | 62 | 38 | 41 | 28

3. Post Hoc Outcome: Comparison of Response Rates of Three Different Doses of HAL PDT and Placebo at 6 Months After First Treatment.
Description: Response was defined as absence of HSIL, and absence of oncogenic HPV if LSIL.
Time Frame: 6 months after first treatment
Population: Patients diagnosed with HSIL histology by a panel of pathologists were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | HAL 5% With Illumination | HAL 1% With Illumination | HAL 0.2% With Illumination | Placebo Ointment Without Illumination
Number analyzed (Participants) | 21 | 22 | 23 | 18
percentage of participants | 76 | 45 | 43 | 28

4. Post Hoc Outcome: Comparison of Response Rates of Three Different Doses of HAL PDT and Placebo at 9 Months After First Treatment
Description: Response was defined as absence of HSIL, and absence of oncogenic HPF if LSIL
Time Frame: 9 months after first treatment
Population: Patients diagnosed with HSIL histology by a panel of pathologists were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | HAL 5% With Illumination | HAL 1% With Illumination | HAL 0.2% With Illumination | Placebo Ointment Without Illumination
Number analyzed (Participants) | 21 | 22 | 23 | 18
percentage of participants | 76 | 50 | 43 | 33

ADVERSE EVENTS:
Arm/Group | HAL 5% With Illumination | HAL 1% With Illumination | HAL 0.2% With Illumination | Placebo Ointment Without Illumination
Serious Adverse Events (participants affected / at risk) | 2/65 | 1/67 | 0/62 | 0/68
Other Adverse Events (participants affected / at risk) | 40/65 | 29/67 | 23/62 | 33/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HAL 5% With Illumination (N=65) | HAL 1% With Illumination (N=67) | HAL 0.2% With Illumination (N=62) | Placebo Ointment Without Illumination (N=68)
Salpingo-oophoritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Adnexitis
Tubo-ovarian abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HAL 5% With Illumination (N=65) | HAL 1% With Illumination (N=67) | HAL 0.2% With Illumination (N=62) | Placebo Ointment Without Illumination (N=68)
Local discomfort (Reproductive system and breast disorders) | 24 (33) | 12 (15) | 9 (9) | 10 (13) — Includes pelvic pain, vulvovaginal discomfort, vulvovaginal burning sensation, vulvovaginal pain, genital pain, uterine cervical pain, uterine spasm, abdominal pain/discomfort, procedural pain, post procedural discomfort
Discharge (Reproductive system and breast disorders) | 22 (27) | 12 (17) | 9 (10) | 8 (9)
Spotting (Reproductive system and breast disorders) | 6 (6) | 8 (8) | 7 (7) | 4 (6) — Includes vaginal haemorrhage, cervix haemorrhage uterine and metrorrhagia
Local infection (Reproductive system and breast disorders) | 6 (9) | 2 (2) | 3 (3) | 9 (10) — Includes vaginal infection, cervicitis, fungal/mycotic infections, vulvitis and trichomonasis
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 2 (3) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less